CLINICAL TRIAL: NCT06764316
Title: A Multicenter, Open Label, Non-randomized First-in-human Phase 1 Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of BAY 3547926 Alone, and in Combination, in Participants With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A First-in-human Study to Learn About the Safety of BAY 3547926 and How Well it Works in Participants With Advanced Liver Cancer
Acronym: BANTAM-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22262; 2024-516615-25-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-12-18; First posted 2025-01-08 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma (HCC); Locally advanced HCC; Metastatic HCC; Unresectable HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BAY 3547926 (Experimental): actinium-225 labeled antibody conjugate
  Interventions: Drug: BAY 3547926; Drug: BAY 3547922

INTERVENTIONS:
Drug: BAY 3547926 — antibody conjugate with actinium-225 label
Drug: BAY 3547922 — antibody conjugate without actinium-225 label as preinjection

SUMMARY:
In this study, researchers want to learn about the safety of a new drug, BAY 3547926, and how well the drug works in people with a type of liver cancer called advanced hepatocellular carcinoma (HCC), which has a special protein called Glypican 3 (GPC3). Researchers want to find the best dose of BAY 3547926 for people with advanced HCC and look at the way the body absorbs and distributes the drug.

The study drug, BAY 3547926, delivers a radioactive agent to cancer cells. The radioactive agent emits radiations which can damage the cancer cells and cause them to die. These radiations travel a small distance, so are expected to cause little damage to surrounding healthy tissues. This is the first study of BAY 3547926 in humans.

Participants will take part in one of the 3 different parts of the study. In Part 1, participants will receive different doses of BAY 3547926 alone to find the dose that is deemed safe and works best for the participants. When this dose has been found, a larger number of participants will receive BAY 3547926 alone in Part 2 or with other treatments in Part 3 of the study.

During the study, the doctors and their study team will do health check-ups, take pictures (scans) of the body, collect blood and urine samples, and ask participants questions about how they are feeling and what health problems they are having.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable HCC (hepatocellular carcinoma) with histological or cytological confirmation, or non-invasive diagnosis as per American Association for the Study of Liver Diseases (AASLD) criteria in participants with a confirmed diagnosis of cirrhosis.
* Demonstrated positive centrally confirmed GPC3 expression by immunohistochemistry (IHC) on tumor sample.
* Disease not amenable to, or progressive disease after, curative surgery and/or locoregional therapies of established efficacy such as resection, local ablation, chemoembolization.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* At least one measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1. as assessed by local site Investigator within 28 days prior to the start of the study treatment.
* Adequate bone marrow and organ function

Exclusion Criteria:

* Fibrolamellar HCC, sarcomatoid HCC, and mixed hepatocellular/cholangiocarcinoma subtypes.
* Participants with a history or clinical evidence of CNS metastases, unless they meet specific criteria
* History of encephalopathy ≥ Grade 2 within the past 12 months
* Clinically significant ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1 (dose escalation): Occurrence and severity of TEAEs | up to 60 months after first administration
  TEAE=Treatment emergent adverse event
Part 1 (dose escalation): Recommended safe and active dose (RSAD) | up to 60 months after first administration
  The RSAD is based on incidence of DLT and preliminary anti-tumor activity (ORR using RECIST 1.1 by Investigator assessment) informed by TITE-CRM.
  RSAD=Recommended safe and active dose DLT=Dose limiting toxicity ORR=Objective reponse rate RECIST=Response Evaluation Criteria in Solid Tumors TITE-CRM =Time-to-event continual reassessment method
Part 2 (dose expansion): Occurrence and severity of TEAEs | up to 60 months after first administration
  TEAE=Treatment emergent adverse event
Part 2 (dose expansion): ORR using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  ORR=Objective reponse rate RECIST=Response Evaluation Criteria in Solid Tumors
Part 2 (dose expansion): DCR using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  DCR=Disease control rate RECIST=Response Evaluation Criteria in Solid Tumors
Part 2 (dose expansion): DoR using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  DoR=Duration of response RECIST=Response Evaluation Criteria in Solid Tumors
Part 2 (dose expansion): PFS using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  PFS=Progression free survival RECIST=Response Evaluation Criteria in Solid Tumors
Part 3 (dose expansion in combination): Occurrence and severity of TEAEs | up to 60 months after first administration
  TEAE=Treatment emergent adverse event
Part 3 (dose expansion in combination): ORR using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  ORR= Objective response rate
Part 3 (dose expansion in combination): DCR using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  DCR=Disease control rate
Part 3 (dose expansion in combination): DoR using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  DoR=Duration of response
Part 3 (dose expansion in combination): PFS using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  PFS=Progression free survivial

SECONDARY OUTCOMES:
Part 1 (dose escalation): Recommended dose level(s) based on occurrence and severity of TEAEs and DLTs, PK, immunogenicity, and preliminary anit-tumor activity (ORR using RECIST 1.1 by Investigator assessment) | up to 60 months after first administration
  TEAE=Treatment emergent adverse event DLT=Dose limiting toxicity PK=Pharmacokinetic ORR=Objective response rate RECIST=Response Evaluation Criteria in Solid Tumors
Part 1 (dose escalation): Recommended dosing regimen based on occurrence and severity of TEAEs and DLTs, PK, immunogenicity, and preliminary anti-tumor activity (ORR using RECIST 1.1 by Investigator assessment) | up to 60 months after first administration
  TEAE=Treatment emergent adverse event DLT=Dose limiting toxicity PK=Pharmacokinetic ORR=Objective response rate RECIST=Response Evaluation Criteria in Solid Tumors
Part 1 (dose escalation): ORR using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  ORR=Objective response rate RECIST=Response Evaluation Criteria in Solid Tumors
Part 1 (dose escalation): DCR using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  DCR=Disease control rate RECIST=Response Evaluation Criteria in Solid Tumors
Part 1 (dose escalation): DoR using RECIST 1.1 by investigator assessment | Up to 60 months after first administration
  DoR=Duration of response RECIST=Response Evaluation Criteria in Solid Tumors
Part 1 (dose escalation): PFS using RECIST 1.1 by investigator assessment | up to 60 months after first administration
  PFS=Progression free survival RECIST=Response Evaluation Criteria in Solid Tumors
Part 1 (dose escalation): Cmax of BAY 3547926 after a single dose and after multiple doses | up to 36 weeks after first administration
  Cmax=Maximal blood concentration
Part 1 (dose escalation): AUC of BAY 3547926 after a single dose and after multiple doses | up to 36 weeks after first administration
  AUC=Area under the blood concentration versus time curve
Part 1 (dose escalation): Clearance of BAY 3547926 after a single dose and after multiple doses if data allow | up to 36 weeks after first administration
  PK=Pharmacokinetic
Part 2 (dose expansion): Recommended dose based on safety, PK, IG and markers of pharmacodynamic activity and efficacy assessments | up to 36 months after first administration
  PK=Pharmacokinetic IG=Immunogenicity
Part 2 (dose expansion): Recommended schedule based on safety, PK, IG and markers of pharmacodynamic activity and efficacy assessments | up to 36 months after first administration
  PK=Pharmacokinetic IG=Immunogenicity
Part 2 (dose expansion): Cmax of BAY 3547926 after a single dose and after multiple doses | up to 36 weeks after first administration
  Cmax=maximal blood concentration
Part 2 (dose expansion): AUC of BAY 3547926 after a single dose and after multiple doses | up to 36 weeks after first administration
  AUC=Area under curve of blood concentration versus time curve
Part 2 (dose expansion): Clearance of BAY 3547926 after single dose and after multiple doses, where applicable and if data allow | up to 36 weeks after first administration
  PK=Pharmacokinetic
Part 3 (dose expansion in combination): Recommended dose level(s) of BAY 3547926 based on clinical data including, but not limited to, occurrence and severity of TEAEs and DLTs, PK and IG | up to 60 months after first administration
  TEAE=Treatment emergent adverse event DLT=Dose limiting toxicity PK=Pharmacokinetic IG=Immunogenicity
Part 3 (dose expansion in combination): Recommended dosing regimen of BAY 3547926 based on clinical data including, but not limited to, occurrence and severity of TEAEs and DLTs, PK and IG | up to 60 months after first administration
  TEAE=Treatment emergent adverse event DLT=Dose limiting toxicity PK=Pharmacokinetic IG=Immunogenicity
Part 3 (dose expansion in combination): Recommended schedule of BAY 3547926 based on severity of TEAEs, PK, IG | up to 60 months after first administration
  TEAE=Treatment emergent adverse event DLT=Dose limiting toxicity PK=Pharmacokinetic IG=Immunogenicity
Part 3 (dose expansion in combination): Cmax of BAY 3547926 after a single dose and after multiple doses of BAY 3547926 in combination | up to 60 months after first administration
  Cmax=maximal blood concentration
Part 3 (dose expansion in combination): AUC of BAY 3547926 after single dose and after multiple doses of BAY 3547926 in combination | up to 60 months after first administration
  AUC=Area under curve of blood concentration versus time curve
Part 3 (dose expansion in combination): Clearance of BAY 3547926 after single dose and after multiple doses of BAY 3547926 in combination, where applicable and if data allow | up to 60 months after first administration
  PK=Pharmacokinetic

CONTACTS AND LOCATIONS:
Locations (10):
- Belgium (2):
  - UZA - Digestive Oncology, Edegem
  - az Groeninge - Digestive Oncology, Kortrijk
- Canada (3):
  - Centre Hospitalier de l'Universite de Montreal (CHUM) - Hopi, Montreal, Quebec
  - McGill University Health Centre (MUHC) - Research Institute (RI) - McConnell Centre for Innovative Medicine (CIM), Montreal, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec
- Finland (2):
  - Tampere University Hospital, Cancer Center, Tampere
  - Turku University Hospital - Oncology Department, Turku
- The START Center for Cancer Care - Madrid - CIOCC - Hospital Universitario Madrid Sanchinarro - Oncologia, Madrid, Spain
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust | Sutton - Gastrointestinal Unit, Sutton, Surrey
  - Imperial College Healthcare NHS Trust | Hammersmith Hospital - Garry Weston Centre, London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.